CLINICAL TRIAL: NCT03985176
Title: Delayed Cerebral Ischaemia and Coagulation Alterations After Aneurysmal Subarachnoid Haemorrhage: a Clinical Observational Trial
Brief Title: Delayed Cerebral Ischaemia and Coagulation Alterations After Aneurysmal Subarachnoid Haemorrhage
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Tampere University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R18110
Record Dates: First submitted 2019-06-05; First posted 2019-06-13 (Actual); Last update posted 2022-11-10 (Actual); Status verified 2022-10

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
Keywords: aneurysmal subarachnoid hemorrhage; delayed cerebral ischemia; Intensive Care Unit; Neurosurgery
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples Without DNA — The total amount of blood collected 109.5 ml
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aneurysmal SAH patients: Patients suffering from aneurysmal subarachnoid haemorrhage
  Interventions: Device: ROTEM; Procedure: EEG; Procedure: bilateral compression ultrasound of the lower extremity veins

INTERVENTIONS:
Device: ROTEM — ROTEM measurements 24,48, 72, 120, 192 and 288 hours from aneurysmal SAH
Procedure: EEG — Continuous EEG-monitoring after aneurysm treatment until patient transferred to ward or up to 14 days after aneurysmal SAH
Procedure: bilateral compression ultrasound of the lower extremity veins — to exclude asymptomatic deep venous thrombosis once over days 3 to 7

SUMMARY:
Despite the advances in neurosurgical and -radiological techniques and intensive care, the mortality and morbidity rates in SAH have not changed in recent years. There is still only a limited understanding of the mechanisms of secondary insults causing brain injury after SAH, also called delayed cerebral ischemia (DCI).

In this study, the investigators are exploring the use of quantifiable biomarkers from blood and continuous EEG monitoring as tools for the diagnostics of DCI. Additionally, the investigators are looking into other clinical variables (eg. pain, heart function) as factors of DCI.

DETAILED DESCRIPTION:
Subarachnoidal hemorrhage (SAH) is a cause of long-term disability and death. Annually about 1000 people in Finland suffer from SAH, their average age being under 50 years. SAH has a mortality rate of 12 % acutely and 40 % of patients die within a month from admission to hospital. In addition, 30 % of the surviving patients remain with neurological deficits. Most survivors of the primary insult suffer from a secondary injury during the first 2-3 weeks from the insult.

Despite the advances in neurosurgical and -radiological techniques and intensive care, the mortality and morbidity rates in SAH have not changed in recent years. There is still only a limited understanding of the mechanisms of secondary insults causing brain injury after SAH, also called delayed cerebral ischemia (DCI).

In this study, the investigators are exploring the use of quantifiable biomarkers from blood and continuous EEG monitoring as tools for the diagnostics of DCI. Additionally, the investigators are looking into other clinical variables (eg. pain, heart function) as factors of DCI.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Admitted to the Tampere University Hospital ICU due to aneurysmal SAH
* Acute subarachnoid haemorrhage (confirmed by computed tomography, CT, AND confirmed origin either with computed angiography (CTA) or digital subtraction angiography (DSA)
* Definite or approximated time for the onset of symptoms and delay to ICU admission no more than 24 hours
* Expected treatment time at least 120 hours in the Tampere University Hospital

Exclusion Criteria:

* Known pregnancy
* Any long-term anticoagulant or antithrombotic medication, except for low-dose aspirin (under 150 mg/day)
* Known active cancer or cirrhotic liver disease or end-stage renal disease requiring renal replacement therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from aneurysmal subarachnoid haemorrhage
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2019-06-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of delayed cerebral ischemia | 14 days
  Incidence of DCI (delayed cerebral ischemia)

SECONDARY OUTCOMES:
Maximal clot firmness of FIBTEM (FIBTEM-MCF) analysis | at 72 hours
  Maximal clot firmness of FIBTEM analysis (FIBTEM-MCF) using rotational thromboelastometry (ROTEM) assay
Incidence of deep venous thrombosis | Within 3-7 days
  Incidence of deep venous thrombosis
Other rotational thromboelastometry analysis | from 24 to 288 hours
  Maximal clot firmness of extrinsic (EXTEM) analysis (EXTEM-MCF) using rotational thromboelastometry
Assessment of neurological outcome | 90 days
  Description of the neurological outcome by using extended Glasgow Outcome Score
  1. Death
  2. Vegetative sate
  3. Lower severe disability
  4. Upper severe disability
  5. Lower moderate disability
  6. Upper moderate disability
  7. Lower good recovery
  8. Upper good recovery
Assessment of pain | Up to 14 days
  Critical Care Pain Observation Tool values, from 0: no pain to 8: maximum pain
Assessment of cardiopulmonary function by transthoracic echocardiography | At admission and at at 24±4 hours
  Function of the left and right ventricle using scale 1. hyperkinetic,2. normal, 3. moderately impaired, 4. severely impaired
Continuous electroencephalography | From 48 hours to 14 days
  Continuous electroencephalography will be evaluated for signs that are potential surrogates of developing delayed cerebral ischemia (such as alpha-delta-ratio, focal slowing, epileptiform abnormalities, relative alpha variability)
Neuroglial brain injury biomarkers | From 24 to 288 hours
  Peripheral blood biomarkers potentially reflecting neuroglial injury will be analysed with enzyme-linked immunosorbent assays

CONTACTS AND LOCATIONS:
Overall Officials: Simo Varila, Study Chair — Tampere University Hospital
Locations (1):
- Tampere University Hospital, Tampere, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Raatikainen E, Kiiski H, Kuitunen A, Junttila E, Huhtala H, Kallonen A, Ala-Peijari M, Langsjo J, Saukkonen J, Valo T, Kauppila T, Raerinne S, Frosen J, Vahtera A. Increased blood coagulation is associated with poor neurological outcome in aneurysmal subarachnoid hemorrhage. J Neurol Sci. 2024 Mar 15;458:122943. doi: 10.1016/j.jns.2024.122943. Epub 2024 Feb 23. PMID 38422781